CLINICAL TRIAL: NCT03614858
Title: Pilot Study of the Efficacy and Safety of Cluster of Differentiation Antigen 19 (CD19) /Cluster of Differentiation Antigen 22 (CD22) CART in the Treatment of Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia.
Brief Title: CD19/CD22-targeted Chimeric Antigen Receptor Engineered T Cell (CART) in B-Cell Acute Lymphoblastic Leukemia.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UnicarTherapy201807
Record Dates: First submitted 2018-07-28; First posted 2018-08-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Leukemia, B-cell
Keywords: CD19; CD22
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Experimental: Cohort 1 Intervention: Biological: CART-19/22 This cohort will determine the safety and efficacy of targeted CD19/CD22 chimeric Antigen Receptor Engineered T Cell Immunotherapy (CART) in the Treatment of CD19/CD22 Positive Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia.
  Interventions: Biological: CART-19/22

INTERVENTIONS:
Biological: CART-19/22 — Split intravenous infusion of CART-19/22 cells of (Dose escalating infusion of 1 - 20 x10^6 CART-19/22 cells/kg).

SUMMARY:
This is a single center, open-label ,phase 1/2 study to evaluate the safety and efficacy of targeted CD19/CD22 chimeric antigen receptor engineered T cell immunotherapy (CART) in the treatment of CD19/CD22 positive Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
The patients will receive infusion of CART cells targeting CD19 and CD22 to confirm the safety and efficacy of CD19/CD22 CART Cells in Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with CD19+/CD22+ relapsed/refractory B-cell acute lymphoblastic leukemia who have a dismal prognosis (estimated survival from several months to <2 year). The study will enroll 20 evaluable patients as follows:
* Age 6-65 years.
* Left ventricular ejection fractions≥ 0.5 by echocardiography.
* Creatinine < 1.6 mg/dL.
* Aspartate aminotransferase/aspartate aminotransferase < 3x upper limit of normal.
* Bilirubin <2.0 mg/dL.
* Karnofsky performance status ≥ 60
* Expected survival time ≥ 3 months (according to investigator's judgement)

Exclusion Criteria:

* Pregnant or lactating women.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification.
* HIV infection.
* Patients with history of seizure
* Active central nervous system leukemia

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months
  Adverse events are evaluated with CTCAE V4.03

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China